CLINICAL TRIAL: NCT06491407
Title: ANALYSIS OF FACTORS INFLUENCING CHEWING AND SWALLOWING PERFORMANCE IN GERIATRICS WITHIN THE SCOPE OF INTERNATIONAL CLASSİFİCATION OF FUNCTIONING, DISABILITY, AND HEALTH
Brief Title: RISK FACTOR ANALYSIS OF CHEWING AND SWALLOWING PERFORMANCE IN GERIATRICS
Status: Recruiting | Type: Observational
Sponsor: Atılım University (Other)
Collaborators: Hacettepe University (Other)
Responsible Party: Principal Investigator, Sena Nur Begen, Research Assistant, Hacettepe University
Other Study IDs: SBA 23/421
Record Dates: First submitted 2024-07-01; First posted 2024-07-09 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Swallowing Disorder; Chewing Problem; Geriatrics
Keywords: swallow; chewing; geriatrics; risk factor
MeSH Terms: conditions — Deglutition Disorders | interventions — Mastication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Geriatrics: >65 years old individuals
  Interventions: Diagnostic Test: Chewing and swallowing performance assessment and related factors

INTERVENTIONS:
Diagnostic Test: Chewing and swallowing performance assessment and related factors — In the study, the dependent variables, chewing performance, will be evaluated with the Chewing and Swallowing Test of Solids, and swallowing performance will be assessed with the Repetitive Saliva Swallowing Test and Dysphagia Limit. Independent variables affecting chewing and swallowing performance have been considered within the scope of the ICF, and all possible factors determined for both geriatrics and swallowing have been listed, and the evaluation parameters and assessment tools have been decided.

SUMMARY:
Various structural and functional problems in neural, sensory and perceptual, cardiovascular, pulmonary, gastrointestinal, endocrine, and musculoskeletal systems occur in geriatrics not associated with a specific disease. One of the problems observed in geriatrics is chewing and swallowing disorders. Failure to detect changes in chewing and swallowing performance in elderly individuals at an early stage may lead to chewing and swallowing disorders and serious complications in later stages. Therefore, it is necessary to comprehensively and systematically address the possible factors affecting chewing and swallowing performance in geriatric individuals.

The first aim of the study is to analyze the factors affecting chewing and swallowing performance in geriatric individuals within the scope of the International Classification of Functioning, Disability, and Health (ICF). The second aim of the study is to create a dysphagia risk prediction model for geriatric individuals based on the results of the analyses to be conducted.

In the study, the dependent variables, chewing performance, will be evaluated with the Chewing and Swallowing Test of Solids, and swallowing performance will be assessed with the Repetitive Saliva Swallowing Test and Dysphagia Limit. Independent variables affecting chewing and swallowing performance have been considered within the scope of the ICF, and all possible factors determined for both geriatrics and swallowing have been listed, and the evaluation parameters and assessment tools have been decided. The evaluation parameters have been categorized under ICF headings such as personal factors, body structures, body functions, activity and participation, and environmental factors, and the evaluations to be conducted have been divided into two groups: geriatric and physiotherapy evaluations. The geriatric evaluations are part of routine geriatric assessment and do not include any specific evaluation for the study. Physiotherapy evaluations will be applied in a certain order to use time efficiently and will take approximately 35-45 minutes. Through geriatric and physiotherapy evaluations, a holistic assessment of participants within the scope of ICF will be ensured.

ELIGIBILITY:
Inclusion Criteria:

* being voluntary to participation,
* Being over 65 years old,
* Understanding and following simple instructions,
* Being able to walk independently for 4 meters.

Exclusion Criteria:

* Having a problem that prevents communication and/or following simple instructions.

Ages: 65 Years to 120 Years | Sex: All
Age Groups: Older Adult
Study Population: Geriatrics over the age of 65 who come for routine examination for Hacettepe University Hospital Geriatri Clinis will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Chewing performance | 1 day
Swallowing performance | 1 day

SECONDARY OUTCOMES:
Deccriptive informations | 1 day
Fragility Assessment | 1 day
posture assessment | 1 day
oral structure assessment | 1 day
cognitive assessment | 1 day
emotional status assessment | 1 day
appetite assessment | 1 day
sleep assessment | 1 day
hearing and vision assessment | 1 day
taste and smell assessment | 1 day
intraoral sensation assessment | 1 day
Temporomandibular pain assessment | 1 day
fonation assessment | 1 day
articulation assessment | 1 day
Respiratory assessment | 1 day
exercise tolerance assessment | 1 day
Feeding and oral intake assessment | 1 day
Laryngeopharyngeal reflux assessment | 1 day
oral health assessment | 1 day
oral dryness assessment | 1 day
swallow problems assessment | 1 day
Temporomandibular joint range of motion | 1 day
jaw openin force | 1 day
hand grip | 1 day
5 repetetion sit to stand test | 1 day
Timed up and go | 1 day
basic functional independance assessment | 1 day
enstrümental functional independance assessment | 1 day
social support assessment | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Selen serel arslan, Prof, Study Director — Hacettepe University
Locations (1):
- Atılım Uiveristy, Ankara, Incek, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No